CLINICAL TRIAL: NCT01833689
Title: Glycaemic Index Testing of Carbohydrate Containing Foods Using a Standardised Method
Brief Title: Glycaemic Index of Foods in Healthy Volunteers
Acronym: GI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13HH0549
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: glucose response; glycaemic index

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- food consumption: control (Placebo Comparator): The control product will be 50g glucose powder dissolved in 250ml of water
  Interventions: Dietary Supplement: food consumption
- food consumption: product (Active Comparator): The test food will provide 50g of available carbohydrate
  Interventions: Dietary Supplement: food consumption

INTERVENTIONS:
Dietary Supplement: food consumption — Reference food The reference food is 50 g glucose powder dissolved in 250ml water
  Test foods The test foods are prepared according to manufacturer's instructions, representing the food as normally consumed. The test foods are consumed once only on separate occasions as a portion providing 50g of available carbohydrate.
  Breakfast cereals should be consumed with 150 ml milk which is additional to the 50 g available carbohydrate in the cereal. In testing breakfast cereals, the reference food must also be consumed with an additional 150 ml milk.

SUMMARY:
The objective of this study is to assess the effect that dietary carbohydrates have on blood sugar by measuring the glycaemic index. The glycaemic index is a comparison between the effect of equal amounts of carbohydrate from a test food compared to a standard (in this case glucose) on blood sugar.

Different foods that contain different carbohydrates have different effects on blood sugars. This is of interest as a number of studies have shown that the level of sugar in the blood after a meal relates directly to the risk of developing heart disease and diabetes. The aim of collecting this data is to be able to give advice to people about the carbohydrates they eat to reduce the risk of diabetes and heart disease.

DETAILED DESCRIPTION:
The study is a randomized cross-over controlled trial: the order of the test foods will be randomized by an independent internet-based program; each participant will be asked to consume all the products; the test food will be compared with a control (in this case 50g glucose).

Suitable subjects will be invited for a screening visit to check for eligibility criteria. Body weight and height measurements will be taken as well as a standard biochemical and haematological screen. If they are eligible and willing to take part, volunteers will be entered into a database and contacted when a GI test becomes available. Volunteers may take part in more than one GI testing up to a maximum of 40 visits per year. Volunteers may withdraw from the database or the study at any time without giving any reason.

Subjects will be asked to come for a set amount of visits for each GI test depending on the number of product that need to be tested (minimum 3 maximum 12 visits for each testing). The volunteers will be informed of the number of visits before they enter the GI testing. For each visit, subjects are tested in the morning after a 10-12h overnight fast.

Three fasting blood samples are taken (-5, -3, -1) 2 minutes apart after which subjects consume the test meal or reference food at an even rate over 15 min. All subjects are asked to record the time it takes in minutes to consume the test food/reference. Further blood samples are taken at 15, 30, 31, 32, 45, 60, 90 and 120 min after the beginning of the meal. The test meal and reference food should be consumed with a 250ml drink of water. This remains constant for each of the tests in the series.

Blood is obtained by finger-pricking using disposable Unistix needles. In previous studies, capillary blood has yielded less between-subject variation in GI. Instant glucose analysers will be used.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-27 kg/m2
* age 18-65 years
* healthy

Exclusion Criteria:

* diabetes
* chronic disease
* glucose impairment
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
glycaemic index | 1-2 months depending on product

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, BSc SRD PhD, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial CRF, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No